CLINICAL TRIAL: NCT05321758
Title: Repeated and Multiple Fecal Microbiota Transplantations Plus Partial Enteral Nutrition as the First-line Treatment in Active Pediatric Crohn's Disease
Brief Title: Fecal Microbiota Transplantation as the First-line Treatment in Active Pediatric Crohn's Disease
Acronym: FMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Biao Zou, attending physician, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83663594
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
Keywords: Crohn Disease;fecal microbiota transplantation
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation; Immunosuppressive Agents

STUDY DESIGN:
Intervention Model Description: Partial enteral nutrition,FMT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT group (Active Comparator): Repeated and multiple FMTs plus PEN(80%) in the treatment of pediatric CD. Patients received PEN (80% of total calories as a polymeric diet, Peptamen, Nestle, Vevey, and Switzerland) and FMT intervention. In the induction stage of CD, FMT was given 1-3 courses, 3-6 times per course.
  Interventions: Biological: Fecal Microbiota Transplantation
- Immunosuppressive group (Sham Comparator): Patients received PEN (80% of total calories as a polymeric diet, Peptamen, Nestle, Vevey, and Switzerland) combined with Immunosuppressants (hormones, azathioprine, thalidomide) treatment.
  Interventions: Drug: Immunosuppressive Agents

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — In the induction stage of CD, FMT was given 1-3 courses, 3-6 times per course.
  Other Names: FMT
  Arms: FMT group
Drug: Immunosuppressive Agents — hormones, azathioprine, thalidomide
  Other Names: Immunosuppressive group
  Arms: Immunosuppressive group

SUMMARY:
To explore the safety and effectiveness of repeated and multiple fecal microbiota transplantations (FMTs) plus partial enteral nutrition (PEN) as a first-line treatment for active Crohn's disease (CD) in children.

DETAILED DESCRIPTION:
Recent studies have suggested that gut imbalance and deregulation of immunological responses plays a pivotal role in the disease development of Crohn's disease (CD), and that FMT could be a useful treatment. Our study is aims to repeated and multiple FMTs plus PEN as a first-line treatment for active Crohn's disease (CD) in children. The patients were divided into 2 groups voluntarily. Patients treated with FMT coupled with PEN were defined as the FMT group, and those treated with PEN combined with Immunosuppressants (hormones, azathioprine, thalidomide) served as the Immunosuppressive group. The therapeutic effect of the two groups was compared. In the induction stage of CD, FMT group received FMT and PEN intervention, and FMT was given 1-3 courses, 3-6 times per course. The transplantation routes include oral capsule, enema and/or colonoscopy. All the patients received PEN (80% of total calories as a polymeric diet, Peptamen, Nestle, Vevey, and Switzerland) intervention to help induce and maintain clinical remission.

ELIGIBILITY:
Inclusion Criteria:

age of older than 2 years and younger than 16 years with no genetic diseases; newly diagnosed with mild-to-moderate CD ( defined by the PCDAI of >10 and ≤40, and SES-CD of >3); Subjects with no change in medication or dose at least 1 week prior to transplantation; agree to received regularly colonoscopy

Exclusion Criteria:

patients who were treated with corticosteroids, methotrexate, thiopurines, and anti-TNF agents as their first-line treatment

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-03-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 8-12 weeks after FMT
  Clinical remission defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score≤10
Endoscopic remission | 8-12 weeks after FMT
  Endoscopic remission defined by a Simple Endoscopic Score for CD （SES-CD) ≤ 2
Mucosal healing | 8-12 weeks after FMT
  Mucosal healing defined as SES-CD = 0

SECONDARY OUTCOMES:
Adverse events | 2 and 10 weeks after FMT
  All possible adverse events:fever,abdominal pain,infectious diseases and others

OTHER OUTCOMES:
gut microbial | before treatment and 5-10 weeks after treatment
  Fecal 16S RNA or macrogene sequencing was performed. Fecal samples were obtained from donor and recipient. The fecal samples and isolated microbiota samples were frozen immediately and underwent DNA extraction using standard methods.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Huang, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zou B, Liu S, Dong C, Shen H, Lv Y, He J, Li X, Ruan M, Huang Z, Shu S. Fecal microbiota transplantation restores gut microbiota diversity in children with active Crohn's disease: a prospective trial. J Transl Med. 2025 Mar 6;23(1):288. doi: 10.1186/s12967-024-05832-1. PMID 40050917